CLINICAL TRIAL: NCT03861091
Title: A Randomized Clinical Trial of Prophylactic Risedronate for Patients With Peripheral Lung Tumors Treated With SBRT
Brief Title: Prophylactic Risedronate for Patients With Peripheral Lung Tumors Treated With SBRT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00056835; CCCWFU99518 (Other: Wake Forest Baptist Comprehensive Cancer Center); P30CA012197 (NIH)
Record Dates: First submitted 2019-02-28; First posted 2019-03-04 (Actual); Results first posted 2023-07-14 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Lung Neoplasm
MeSH Terms: conditions — Lung Neoplasms | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Risedronate (Experimental): Risedronate 150 mg given once 7-21 days prior to initiation of SBRT
  Interventions: Drug: risedronate
- Matching Placebo (Placebo Comparator): Matching placebo, dose not applicable given once 7-21 days prior to initiation of SBRT
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: risedronate — Risedronate 150 mg Oral Given once 7 - 21 days prior to initiation of SBRT
  Other Names: Actonel; Atelvia
  Arms: Risedronate
Drug: Matching placebo — Dose not applicable, given once 7-21 days prior to initiation of SBRT
  Arms: Matching Placebo

SUMMARY:
This is a double blind randomized controlled study investigating the efficacy of a single dose of 150 mg risedronate (a bone anti-resorptive) vs a single dose of placebo given prior to SBRT for peripheral lung tumors that are within 2 cm of the chest wall. Our hypothesis is that the use of a single dose of 150 mg risedronate will eliminate or greatly reduce the rapid bone loss that occurs with radiation induced early osteoclast recruitment/activation.

Patients will be given either a single dose of 150 mg risedronate or placebo at the time of their treatment mapping "simulation" CT scan. Typically, radiation treatments begin at 1 - 3 weeks following this mapping scan, as each treatment plan requires detailed physics calculations and quality assurance checks.

All CT imaging referenced below is performed as a routine standard of care surveillance and is necessary for cancer treatment follow-up. These chest CT scans that are utilized in this research protocol would be performed every 3 months regardless of inclusion on this trial.

DETAILED DESCRIPTION:
2.1 Primary Objective(s)

The primary objective is to assess the percent change in bone mean cortical thickness within regions of bone receiving 30 Gy or more at 3 months after SBRT. The % change in mean cortical thickness will be compared between patients who received risedronate and those who received placebo.

2.2 Secondary Objective(s)

In addition to the primary objective, the investigators will further analyze the remaining routine follow-up chest CT scans, for mean cortical thickness change in regions of bone that received 0 - 10 Gy, >10 - 20 Gy, > 20 - 30 Gy, > 30 - 40 Gy, and > 40 Gy at all time points including 3 months, 6 months, 9 months, and 12 months. These scans are standard of care and would be performed regardless of inclusion on this trial. This will allow us to determine the potential persistence of effects from SBRT and bisphosphonate use.

The investigators will assess and compare the incidence and grade (per modified CTCAE v.5) of radiation induced chest wall pain within the radiation treatment portal (within the 50% isodose line) at time of each routine follow up visit (3 months, 6 months, 9 months, and 12 months post SBRT). The purpose of utilizing a placebo and double-blind design is that chest wall pain is a subjective finding. Furthermore, it is unclear if chest wall pain from radiation is directly due to bone damage, nerve damage, muscle irritation, or a combination of all of these factors. The use of placebo will help us reduce the potential for bias in pain assessment.

The investigators will assess and compare the incidence of rib and vertebral fractures (as noted on CT imaging) that occur within 12 months of irradiation and are within the radiation treatment field. The radiation treatment field will be defined as within the 50% isodose line.

The urine concentration of an osteoclast-specific biomarker, urinary N-telopeptide (NTX) indicating osteoclast activity will be assessed prior to SBRT and at each routine follow up visit (at 3 months, 6 months, 9 months, and 12 months post SBRT).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years or older, but there is no upper limit on age of inclusion.
* Patients must have a peripheral lung tumor that is amenable to SBRT as determined by the treating radiation oncologist. To be classified as a peripheral lung tumor, the tumor edge (the edge of the gross tumor volume or GTV in radiation treatment planning software) must be within 2 cm of the chest wall. This is determined by the treating radiation oncologist. The chest wall is defined as the chest wall musculature or ribs/vertebrae immediately adjacent to the lungs.
* Patients must have ECOG status of 0-3
* Patients must have a life expectancy of at least 3 months as determined by the treating radiation oncologist.
* Patients must have the ability to understand and the willingness to sign an IRB-approved informed consent document.

Exclusion Criteria:

Prior radiation to any part of the body including the lungs or thorax is not an exclusion criteria

* Tumor edge is greater than 2 cm from the chest wall. The edge of tumor is the edge of the gross tumor volume or GTV as defined in radiation treatment planning software. This is determined by the treating radiation oncologist.
* Tumors that are expected to require more than 10 fractions of radiation as determined by the treating radiation oncologist.
* History of using bone anti-resorptive agents including bisphosphonates or RANK-L inhibitors within the last 1 year.
* Inability to stand or sit upright for at least 30 minutes, which is necessary for ingestion of risedronate.
* Hypocalcemia defined as serum total calcium lower than 8.5 mg/dL on most recent bloodwork that is within 3 months of administration of study drug/placebo.
* Severe renal impairment (EGFR <30 mL/min) on most recent bloodwork that is within 3 months of administration of study drug/placebo.
* Known allergy to risedronate or other bisphosphonates
* Surgery affecting the bone or dental operations within the last 6 months. This will be explicitly asked and documented in the EMR by treating radiation oncologist.
* Dental operations do not include routine cleaning or cavity fillings
* Dental operations that exclude patients refer to any manipulation of mandible.
* Positive urine pregnancy test in women of child bearing potential within 1 week of registration. Pregnant women are excluded from this study because radiation has clear teratogenic and potentially abortifacient risks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-07-12 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Farris, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - High Point Regional Medical Center, High Point, North Carolina
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Risedronate | Matching Placebo
Started | 41 | 43
Completed | 41 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Risedronate | Matching Placebo | Total
Number analyzed (Participants) | 41 | 43 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.4 (7.9) | 71.1 (7.3) | 71.2 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 25 | 25 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 39 | 43 | 82
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 37 | 39 | 76
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 41 | 43 | 84

OUTCOME MEASURES:

1. Primary Outcome: Changes in Mean Cortical Thickness
Description: The primary outcome measure is the percent change in mean cortical thickness (C.Th) of bones receiving 30 Gy or more at 3 months post SBRT, when compared to pre-SBRT cortical thickness
Time Frame: At baseline and at 3 months post radiation
Population: A small number of participants who were enrolled were not able to have cortical thickness determined at 3 months.
Measure: Mean (Standard Error); unit: percent change in mm cortical thickne
Units Other Than Participants: Bones
Arm/Group | Risedronate | Matching Placebo
Number analyzed (Participants) | 39 | 40
Number analyzed (Bones) | 39 | 40
percent change in mm cortical thickne | 4.24 (3.04) | 7.14 (2.93)

2. Secondary Outcome: 4 Time Points Assessing Change in Mean Cortical Thickness of Bones
Description: The percent change in mean C.Th of bones will be assessed in regions of bone that received 0 - 10 Gy, >10 - 20 Gy, > 20 - 30 Gy, > 30 - 40 Gy, and > 40 Gy at all time points including 3 months, 6 months, 9 months, and 12 months.
Time Frame: At baseline, 3 months, 6 months, 9 months and 12 months post radiation
Population: A small number of participants did not have follow-up cortical thickness measures.
Measure: Mean (Standard Error); unit: percent change in mm cortical thickness
Units Other Than Participants: Bones
Arm/Group | Risedronate | Matching Placebo
Number analyzed (Participants) | 39 | 40
Number analyzed (Bones) | 39 | 40
percent change in mm cortical thickness
  % change cort thickness in region <10 Gy--time 3mo to bl | 13.04 (2.56) | 5.57 (2.50)
  % change cort thickness in region <10 Gy--time 6mo to bl | 10.37 (2.63) | 5.76 (2.57)
  % change cort thickness in region <10 Gy--time 9mo to bl | 12.10 (2.71) | 8.07 (2.59)
  % change cort thickness in region <10 Gy--time 12mo to bl | 11.58 (2.89) | 9.42 (2.70)
  % change cort thickness in region 10-20 Gy--time 3mo to bl | 9.27 (2.78) | 4.97 (2.72)
  % change cort thickness in region 10-20 Gy--time 6mo to bl | 6.24 (2.86) | 3.95 (2.82)
  % change cort thickness in region 10-20 Gy--time 9mo to bl | 7.71 (2.95) | 5.65 (2.82)
  % change cort thickness in region 10-20 Gy--time 12mo to bl | 10.11 (3.14) | 7.30 (2.94)
  % change cort thickness in region 20-30 Gy--time 3mo to bl | 8.40 (2.99) | 3.70 (2.87)
  % change cort thickness in region 20-30 Gy--time 6mo to bl | 5.41 (3.08) | 0.10 (2.95)
  % change cort thickness in region 20-30 Gy--time 9mo to bl | 6.48 (3.18) | 4.94 (2.95)
  % change cort thickness in region 20-30 Gy--time12mo to bl | 7.42 (3.36) | 7.23 (3.08)
  % change cort thickness in region 30-40 Gy--time 3mo to bl | 4.90 (3.22) | 5.20 (3.10)
  % change cort thickness in region 30-40 Gy--time 6mo to bl | 1.98 (3.31) | 3.21 (3.19)
  % change cort thickness in region 30-40 Gy--time 9mo to bl | 3.70 (3.43) | 9.64 (3.19)
  % change cort thickness in region 30-40 Gy--time12mo to bl | 2.23 (3.62) | 11.77 (3.32)
  % change cort thickness in region >30 Gy--time 3mo to bl | 4.24 (3.04) | 7.14 (2.93)
  % change cort thickness in region >30 Gy--time 6mo to bl | 1.66 (3.13) | 6.11 (3.01)
  % change cort thickness in region >30 Gy--time 9mo to bl | 2.12 (3.24) | 10.32 (3.02)
  % change cort thickness in region >30 Gy--time 12mo to bl | -0.42 (3.42) | 11.72 (3.14)
  % change cort thickness in region >40 Gy--time 3mo to bl | 5.83 (8.10) | 12.82 (7.53)
  % change cort thickness in region >40 Gy--time 6mo to bl | 5.62 (8.41) | 20.30 (7.68)
  % change cort thickness in region >40 Gy--time 9mo to bl | 6.03 (8.53) | 21.37 (7.69)
  % change cort thickness in region >40 Gy--time 12mo to bl | -1.44 (8.92) | 17.17 (8.25)

3. Secondary Outcome: Number of Participants With Chest Wall Pain
Description: Chest wall pain incidence and grade will be collected as per modified CTCAE v. 5 within the within the 50% isodose line. Appendix K. Below we report numbers with any chest wall pain of grades 3+ over the year of followup.
Time Frame: At baseline, 3 months, 6 months, 9 months and 12 months post radiation
Population: Some participants did not have sufficient self-reported symptom pain data to determine if, over course of 12 months, they had any chest wall pain of grade 3 or higher
Measure: Count of Participants; unit: Participants
Arm/Group | Risedronate | Matching Placebo
Number analyzed (Participants) | 22 | 28
Participants | 2 | 4

4. Secondary Outcome: Number of Participants With Rib and Vertebral Fracture
Description: Incidence of rib and vertebral fractures (as noted on CT imaging) that occur within 12 months of irradiation and are within the within 50% isodose line.
Time Frame: At 12 months post radiation
Population: For a small number of participants it was not possible to determine clearly if a fracture had occurred within 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Risedronate | Matching Placebo
Number analyzed (Participants) | 38 | 39
Participants | 15 | 11

5. Secondary Outcome: Urine Concentration at 4 Time Points
Description: The urine concentration of an osteoclast-specific biomarker, urinary N-telopeptide (U-NTX) indicating osteoclastic activity will be assessed prior to SBRT and at each routine follow up visit (at 3 months, 6 months, 9 months, and 12 months post SBRT).
Time Frame: At 3 months, 6 months, 9 months and 12 months post radiation
Population: A small number of participants did not have urine samples analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Risedronate | Matching Placebo
Number analyzed (Participants) | 38 | 41
pg/mL
  Urinary NTX values at BL | 499.3 (592.0) | 524.9 (399.4)
  Urinary NTX values at 3mo | 460.2 (514.1) | 494.5 (342.4)
  Urinary NTX values at 6mo | 669.9 (955.9) | 350.7 (301.8)
  Urinary NTX values at 9mo | 536.1 (460.0) | 507.0 (492.2)
  Urinary NTX values at 12mo | 611.0 (494.7) | 411.7 (314.0)

ADVERSE EVENTS:
Time Frame: 30 days from the end of all treatments of radiation, up to 12 months.
Arm/Group | Risedronate | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 1/43
Serious Adverse Events (participants affected / at risk) | 0/41 | 2/43
Other Adverse Events (participants affected / at risk) | 5/41 | 0/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risedronate (N=41) | Matching Placebo (N=43)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorders (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Risedronate (N=41) | Matching Placebo (N=43)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/91/NCT03861091/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT03861091/ICF_001.pdf